CLINICAL TRIAL: NCT02914379
Title: Disposition of [¹⁴C]-LY3337641 Following Oral Administration in Healthy Male Subjects
Brief Title: A Study of LY3337641 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16297; I8K-MC-JPDE (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-09-21; First posted 2016-09-26 (Estimated); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2022-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 20mg [¹⁴C]-LY3337641 (Experimental): Participants received 20 milligrams (mg) oral dose of LY3337641 containing 120 microcuries of radioactivity.
  Interventions: Drug: [¹⁴C]-LY3337641

INTERVENTIONS:
Drug: [¹⁴C]-LY3337641 — Administered orally

SUMMARY:
The purpose of this study is to measure how much LY3337641 gets into the bloodstream and how long it takes the body to get rid of it. In addition, the safety and tolerability of the study drug will be evaluated.

Participants will be admitted to a clinical research unit (CRU) the day before dosing. Participants remain confined to the CRU for at least 7 days. Participants may be discharged from the CRU any time after 7 days post-dose (Day 8), and up to a maximum of 21 days post-dose (Day 22).

This study will last approximately 30 days for each participant, not including screening. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males, as determined by medical history and physical examination
* Have a body mass index (BMI) between 18.5 and 32.0 kilograms per meter squared (kg/m²)
* Have clinical laboratory test results within normal reference range for the population or investigative site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling as per the protocol
* Are able and willing to give signed informed consent
* Generally have a minimum of 1 bowel movement per day

Exclusion Criteria:

* Have participated, within the last 30 days, in a clinical trial involving an investigational product. If the previous investigational product has a long half-life, 3 months or 5 half-lives (whichever is longer, if known) should have passed
* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI) (cholecystectomy not acceptable), endocrine, hematological, dermatologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have used or intend to use over-the-counter or prescription medication, including herbal medications, within 14 days prior to dosing
* Have donated blood of more than 500 milliliter (mL) within the month prior to screening
* Have an average weekly alcohol intake that exceeds 21 units per week, and are unwilling to stop alcohol consumption for 48 hours prior to admission, and while resident in the clinical research unit (CRU)
* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study
* Have had exposure to significant diagnostic, therapeutic, or employment related radiation within 12 months prior to dosing (serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring)
* Have participated in a [¹⁴C] study within the last 6 months prior to admission for this study. The total 12-month exposure from this study and a maximum of one other previous [¹⁴C]-study within 6 to 12 months of this study must be within the Code of Federal Regulations (CFR) recommended levels considered safe (per 21 CFR 361.1): less than 5000 Milli-rem (mrem) /year whole body annual exposure

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 20mg [¹⁴C]-LY3337641
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 20mg [¹⁴C]-LY3337641: Participants received 20 mg oral dose of LY3337641 containing 120 microcuries of radioactivity.
Arm/Group | 20mg [¹⁴C]-LY3337641
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Urinary Excretion of Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Description: Urinary excretion samples from each participant were measured by liquid scintillation counting. The radioactive counts detected in urine samples were each divided by the theoretical radioactive count in the total radioactive dose administered and multiplied by 100% to arrive at a percentage of total radioactive dose excreted in urine and feces.
Time Frame: Baseline up to 22 days
Population: All participants who received the study drug and have evaluable pharmacokinetic (PK) data.
Measure: Mean (Standard Deviation); unit: Percentage of total dose
Groups:
- 20 mg [¹⁴C]-LY3337641: Participants received 20 mg oral dose of LY3337641 containing 120 microcuries of radioactivity.
Arm/Group | 20 mg [¹⁴C]-LY3337641
Number analyzed (Participants) | 6
Percentage of total dose | 2.9 (1.0)

2. Primary Outcome: Fecal Excretion of Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Description: Fecal excretion samples from each participant were measured by liquid scintillation counting. The radioactive counts detected in fecal samples were each divided by the theoretical radioactive count in the total radioactive dose administered and multiplied by 100% to arrive at a percentage of total radioactive dose excreted in feces.
Time Frame: Baseline up to 22 days
Population: All participants who received the study drug and have evaluable PK data.
Measure: Mean (Standard Deviation); unit: Percentage of total dose
Arm/Group | 20 mg [¹⁴C]-LY3337641
Number analyzed (Participants) | 6
Percentage of total dose | 86.4 (5.1)

3. Secondary Outcome: Pharmacokinetics: Maximum Observed Concentration (Cmax) of Plasma LY3337641
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264 and 312 hours post dose
Population: All participants who received the study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter (ng/mL)
Arm/Group | 20 mg [¹⁴C]-LY3337641
Number analyzed (Participants) | 6
Nanograms/milliliter (ng/mL) | 77.9 (26)

4. Secondary Outcome: Pharmacokinetics: Maximum Observed Concentration (Cmax) of Plasma Radioactivity
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264 and 312 hours post dose
Population: All participants who received the study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalents/g (ng-equiv/g)
Arm/Group | 20 mg [¹⁴C]-LY3337641
Number analyzed (Participants) | 6
nanogram equivalents/g (ng-equiv/g) | 122 (25)

5. Secondary Outcome: Pharmacokinetics: Maximum Observed Concentration (Cmax) of Whole Blood Radioactivity
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264 and 312 hours post dose
Population: All participants who received the study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 20 mg [¹⁴C]-LY3337641
Number analyzed (Participants) | 6
ng/mL | 67.5 (24)

6. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC 0 to ∞) of Plasma LY3337641
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264 and 312 hours post dose
Population: All participants who received the study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hours per milliliter (ng*h/mL)
Arm/Group | 20 mg [¹⁴C]-LY3337641
Number analyzed (Participants) | 6
Nanograms*hours per milliliter (ng*h/mL) | 370 (25)

7. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC 0 to ∞) of Plasma Radioactivity
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264 and 312 hours post dose
Population: All participants who received the study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng-equivalents*h/gram (ng-equiv*h/g)
Arm/Group | 20 mg [¹⁴C]-LY3337641
Number analyzed (Participants) | 6
ng-equivalents*h/gram (ng-equiv*h/g) | 1240 (51)

8. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC 0 to ∞) of Whole Blood Radioactivity
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264 and 312 hours post dose
Population: All participants who received the study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 20 mg [¹⁴C]-LY3337641
Number analyzed (Participants) | 6
ng*h/mL | 5840 (105)

9. Secondary Outcome: Pharmacokinetics: Total Number of Measurable Metabolites of LY3337641 in Plasma, Urine and Feces
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264, and 312 hours postdose
Population: All participants who received the study drug and have evaluable PK data.
Measure: Number; unit: Number of Metabolites
Arm/Group | 20 mg [¹⁴C]-LY3337641
Number analyzed (Participants) | 6
Number of Metabolites
  Plasma | 6
  Urine | 4
  Feces | 8

ADVERSE EVENTS:
Time Frame: From Baseline to End of Study (Up to 29 Days)
Arm/Group | 20 mg [¹⁴C]-LY3337641
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg [¹⁴C]-LY3337641 (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Change of bowel habit (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days